CLINICAL TRIAL: NCT03355066
Title: A Phase 1, Open-Label, Dose-Escalation, Dose-Finding Study Evaluating the Safety and Pharmacokinetics of Orally Administered SM08502 in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluating the Safety and Pharmacokinetics of Orally Administered SM08502 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due business reasons by Sponsor.
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SM08502-ONC-01
Record Dates: First submitted 2017-11-17; First posted 2017-11-28 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor, Adult
Keywords: SM08502; pan Clk/Dyrk inhibitor; HRR; HRD; LOH High; AR-V7

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A: Dose Escalation (Experimental): Cohorts of subjects with advanced solid tumors will receive increasing doses (10, 20, 40, 60, 80, 120, 160, or 200 mg) of SM08502, administered orally, once daily, following 28-day treatment cycles. If the maximum tolerated dose (MTD) is not determined at the 200 mg dose, dosing will continue at 50 mg/dose increments until an MTD is determined. Cohorts will include approximately 1 to 6 subjects according to an accelerated escalation design and safety requirements for expansion of subject numbers. For the purpose of dose escalation and de-escalation, the dose of SM08502 and regimen may be modified based on the type of dose limiting toxicities (DLTs) observed and following data review and discussions between the Sponsor and Investigators.
  Interventions: Drug: SM08502
- Part 1B: Dose Finding (Experimental): Indications eligible for Part 1B include castration-resistant prostate cancer (CRPC), non-small cell lung cancer (NSCLC), triple-negative breast cancer (TNBC), colorectal cancer (CRC), endometrial cancer, or ovarian cancer for which histologic or cytologic confirmation of malignancy was obtained at diagnosis. Initially, two cohorts of 6-24 subjects will be evaluated comparing 2 different doses and schedules of SM08502 (30 mg daily and 40 mg 5 days on and 2 days off), administered orally following 28-day treatment cycles. If appropriate, alternative doses and schedules may be evaluated depending on the results.
  Interventions: Drug: SM08502
- Part 2: Expansion (Experimental): Part 2 will evaluate the recommended Part 2 dose and schedule of SM08502, as determined in Part 1B, in 3 cohorts of subjects. The indications to be evaluated include subjects with advanced and/or metastatic CRPC (two biomarker selection cohorts) and NSCLC for which histologic or cytologic confirmation of malignancy was obtained at diagnosis. Each cohort will enroll up to 20 subjects.
  Approximately 10 subjects of the total enrolled in Part 2, irrespective of cohort, will be included in a food-effect substudy to assess the preliminary effect of a high-fat, high-calorie meal on the PK of SM08502.
  Interventions: Drug: SM08502

INTERVENTIONS:
Drug: SM08502 — SM08502 tablets to be administered orally.

SUMMARY:
This study is an open-label, multi-center, dose-escalation, dose-finding and expansion study in adult subjects with advanced solid tumors for whom no standard therapy is available. The study will evaluate the safety, tolerability, PK, PD, and preliminary anti-tumor efficacy of SM08502 administered orally, once daily, following a 28-day treatment cycle (Part 1A). Alternative dosing schedules will be explored in Part 1B and the recommended Part 2 dose and schedule will be further evaluated in Part 2.

Subjects will participate in a screening period of up to 14 days. Dosing in 28-day cycles will continue within each subject, unless treatment is discontinued due to toxicity, disease progression, initiation of a new anti-neoplastic therapy, withdrawal of consent, the Sponsor terminates the study, or the subject no longer meets retreatment criteria.

Approximately 10 subjects enrolled in Part 2, irrespective of the tumor type, will be included in a food effect substudy to assess the preliminary effect of a high-fat, high-calorie meal on the PK of SM08502. Subjects participating in the food effect substudy will continue on study and complete assessments as per the Part 2 schedule and receive SM08502 at the recommended Part 2 dose (or another previously assessed dose level and schedule).

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects with advanced solid tumors (as defined below):

   1. Part 1A - Subjects with advanced solid tumors who are refractory to or intolerant of established therapy known to provide clinical benefit for their condition (i.e., subjects must not be candidates for regimens known to provide clinical benefit) and for which histologic or cytologic confirmation of malignancy was obtained at diagnosis, with the exception of hepatocellular carcinoma if it meets appropriate imaging-only diagnostic criteria (per the National Comprehensive Cancer Network [NCCN], Liver Imaging Reporting and Data System [LI-RADS], American Association for the Study of Liver Diseases [AASLD], Asian Pacific Association for the Study of the Liver [APASL], or European Association for the Study of the Liver - European Organisation for Research and Treatment of Cancer [EASL-EORTC]).
   2. Part 1B - Subjects with advanced and/or metastatic solid tumors who are refractory to or intolerant of established therapy known to provide clinical benefit for their condition (i.e., subjects must not be candidates for regimens known to provide clinical benefit in the Investigator's judgment). Histologic or cytologic confirmation of malignancy must have been obtained at diagnosis. The tumor types include: i. NSCLC (adenocarcinoma subtype) ii. TNBC iii. CRPC iv. CRC v. Endometrial cancer (endometrioid subtype) vi. Ovarian cancer (serous, mucinous, and endometrioid subtypes).
   3. Part 2 - Subjects with advanced and/or metastatic solid tumors who are refractory to or intolerant of established therapy known to provide clinical benefit for their condition. Histologic or cytologic confirmation of malignancy must have been obtained at diagnosis. Subjects must have received no more than 2 prior lines of myelosuppressive chemotherapy. Additionally, CRPC subjects must have received no more than 4 total lines of treatment (including any hormonal therapies) in any setting. The tumor types include: i. NSCLC (adenocarcinoma subtype) ii. CRPC in two biomarker selected cohorts.
2. Measurable or evaluable disease per RECIST 1.1 (Part 1A). For Parts 1B and 2, at least 1 measurable lesion per RECIST 1.1 that has not been previously irradiated. In CRPC subjects (Parts 1B and 2) without measurable disease per RECIST 1.1, a PSA that is concordant with clinical disease progression (rising) is eligible. A PSA value of 2 ng/ml or greater is required for study entry.
3. Subjects must have archived tumor specimens available for analysis (as specified in Section 7.2.2). Otherwise, a fresh tumor biopsy will be required at study entry. At the discretion of the Sponsor's Medical Monitor, a fresh tumor biopsy may not be required for eligibility if there are extenuating circumstances (e.g., inaccessible sites of disease or lack of subject suitability to undergo a fresh biopsy, or molecular profiling of archived tissue already performed).
4. Subjects must have recovered (i.e., Grade 1 [or better] based on CTCAE v5.0) from all toxicity associated with previous chemotherapy, targeted therapy, experimental therapy, biological therapy, immuno-oncology therapy, surgery, radiotherapy, or other locoregional therapy (Exceptions include subjects with: continuing alopecia regardless of any CTCAE grade, Grade 2 or lower neuropathy, and well-controlled hypothyroidism and/or adrenal insufficiency on chronic hormone replacement. All subjects with these exceptions are eligible).
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.

Key Exclusion Criteria:

1. Women who are pregnant or lactating
2. Women of childbearing potential (WOCBP) who do not agree to follow the contraceptive guidelines as outlined in the study protocol
3. Men of reproductive potential who do not agree to follow the contraceptive guidelines as outlined in the study protocol
4. Subjects with a corrected QT interval (QTc) using Fridericia's formula (QTcF) > CTCAE v5.0 Grade 1 (>480 msec) based on the mean of triplicate evaluation at Screening.
5. Subjects with clinically significant ventricular tachycardia (VT), atrial fibrillation (AF), ventricular fibrillation (VF), second or third degree heart block
6. Subjects with myocardial infarction (MI) within 1 year, Class II-IV congestive heart failure (CHF) per New York Heart Association (NYHA) classification, or clinically significant coronary artery disease (CAD)
7. Subjects with active infection requiring parenteral antibiotic therapy.
8. Organ transplant recipients.
9. Subjects with known osteoporosis.
10. Subjects with a second malignancy unless adequately treated with no recurrence for 3 years. Subjects with history of previous or recent adequately treated skin basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of any source are eligible.
11. Subjects with active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of SM08502 per Investigator's opinion
12. Subjects with known active human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection
13. Subjects with chronic liver disease or dysfunction and a Child-Pugh score of B or C
14. Subjects with untreated, progressing, or known symptomatic brain metastasis
15. Subjects with retinal abnormalities, specifically diabetic retinopathy, macular degeneration, other forms of retinal degenerative disease, or other retinal findings that may place the subject at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Part 1A, Part 1B: Maximum tolerated dose (MTD) of SM08502 based on the frequency and severity of dose-limiting toxicities (DLTs) | DLT period of 28 days per dose level
Part 1A, Part 1B and Part 2: Number of participants with treatment-emergent adverse events (TEAEs) as assessed by CTCAE v5.0 | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in blood chemistry parameters: blood urea nitrogen [BUN], creatinine, glucose, potassium, sodium, calcium (micromoles per liter) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in blood chemistry parameters: aspartate aminotransferase [AST], alanine aminotransferase (ALT), alkaline phosphatase [ALP] (international units per liter) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in blood chemistry parameters: albumin (grams per day) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in blood chemistry parameters: chloride, bicarbonate (millimoles per liter) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in blood chemistry parameter: lactic acid dehydrogenase [LDH] (units per liter) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in hematology parameter: hemoglobin [Hb] (grams per liter) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in hematology parameter: hematocrit (proportion of red blood cells in blood) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in hematology parameter: red blood cells [RBC] count (trillion cells per liter) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in hematology parameters: neutrophils, lymphocytes, monocytes, eosinophils, basophils, platelet count (cells/microliter) | Approximately 5 years
Part 1A: Change from baseline in prothrombin time [PT] (seconds) | Approximately 5 years
Part 1A: Change from baseline in partial thromboplastin time [PTT] (seconds) | Approximately 5 years
Part 1A: Change from baseline in urinalysis parameter: clarity | Approximately 5 years
Part 1A: Change from baseline in urinalysis parameter: specific gravity (ratio) | Approximately 5 years
Part 1A: Change from baseline in urinalysis parameter: urine pH | Approximately 5 years
Part 1A: Change from baseline in urinalysis parameter: protein | Approximately 5 years
Part 1A: Change from baseline in urinalysis parameter: glucose (millimole per liter) | Approximately 5 years
Part 1A: Change from baseline in urinalysis parameter: ketones (millimoles per liter) | Approximately 5 years
Part 1A: Change from baseline in urinalysis parameter: occult blood (10^9 cells per liter) | Approximately 5 years
Part 1A: Change from baseline in urinalysis parameter: nitrite | Approximately 5 years
Part 1A: Change from baseline in urinalysis parameter: leukocytes (counts per high power field) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in body temperature (degrees celsius) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in pulse rate (beats per minute) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in respiratory rate (breaths per minute) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in blood pressure (systolic and diastolic) (millimeters of mercury) | Approximately 5 years
Part 1A, Part 1B and Part 2: Change from baseline in electrocardiogram (ECG) parameters: PR interval, QRS interval, QT interval, QTcF (milliseconds) | Approximately 5 years
Part 1A and Part 1B: Cmax of SM08502 and its metabolite (SM08955) following single dose administration of SM08502 | Approximately 5 years
Part 1A and Part 1B: tmax of SM08502 and SM08955 following single dose administration of SM08502 | Approximately 5 years
Part 1A and Part 1B: AUC0-24 of SM08502 and SM08955 following single dose administration of SM08502 | Approximately 5 years
Part 1A and Part 1B: AUClast of SM08502 and SM08955 following single dose administration of SM08502 | Approximately 5 years
Part 1A and Part 1B: Cmax,ss of SM08502 and SM08955 following repeat dose administration of SM08502 | Approximately 5 years
Part 1A and Part 1B: Cmin,ss of SM08502 and SM08955 following repeat dose administration of SM08502 | Approximately 5 years
Part 1A and Part 1B: tmax,ss of SM08502 and SM08955 following repeat dose administration of SM08502 | Approximately 5 years
Part 1A and Part 1B: AUC0-24,ss of SM08502 and SM08955 following repeat dose administration of SM08502 | Approximately 5 years
Part 2: Tumor response as measured by RECIST 1.1 (Response Evaluation Criteria In Solid Tumors) or PCWG3 (Prostate Cancer Working Group 3) criteria where appropriate | Approximately 5 years

SECONDARY OUTCOMES:
Part 1A and Part 1B: Tumor response as measured by RECIST 1.1 or PCWG3 criteria where appropriate | Approximately 5 years
Part 1A, Part 1B and Part 2: Gene expression profile of RNA isolated from whole blood | Approximately 5 years
Part 2: Cmax of SM08502 and SM08955 following single dose administration of SM08502 | Approximately 5 years
Part 2: tmax of SM08502 and SM08955 following single dose administration of SM08502 | Approximately 5 years
Part 2: AUC0-24 of SM08502 and SM08955 following single dose administration of SM08502 | Approximately 5 years
Part 2: AUClast of SM08502 and SM08955 following single dose administration of SM08502 | Approximately 5 years
Part 2: Cmax,ss of SM08502 and SM08955 following repeat dose administration of SM08502 | Approximately 5 years
Part 2: Cmin,ss of SM08502 and SM08955 following repeat dose administration of SM08502 | Approximately 5 years
Part 2: tmax,ss of SM08502 and SM08955 following repeat dose administration of SM08502 | Approximately 5 years
Part 2: AUC0-24,ss of SM08502 and SM08955 following repeat dose administration of SM08502 | Approximately 5 years
Part 2: Gene expression and splicing alterations in post-treatment compared to pre-treatment tumor specimens | Approximately 5 years
Part 2 Food Effect substudy: Cmax of SM08502 and SM08955 following single dose administration of SM08502 in fed and fasted states. | Approximately 5 years
Part 2 Food effect substudy: tmax of SM08502 and SM08955 following single dose administration of SM08502 in fed and fasted states. | Approximately 5 years
Part 2: AUC0-24 of SM08502 and SM08955 following single dose administration of SM08502 in fed and fasted states. | Approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Darrin Beaupre, MD, PhD, CMO, Study Chair — Biosplice Therapeutics, Inc.
Locations (19):
- United States (19):
  - Honor Health Research Institute, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope Medical Center, Duarte, California
  - UC Davis - Comprehensive Cancer Center, Sacramento, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Northside Hospital, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - University of Oklahoma Medicine Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - UT Health San Antonio - Mays Cancer Center, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moroney MR, Woodruff E, Qamar L, Bradford AP, Wolsky R, Bitler BG, Corr BR. Inhibiting Wnt/beta-catenin in CTNNB1-mutated endometrial cancer. Mol Carcinog. 2021 Aug;60(8):511-523. doi: 10.1002/mc.23308. Epub 2021 May 26. PMID 34038589
- [Derived] Tam BY, Chiu K, Chung H, Bossard C, Nguyen JD, Creger E, Eastman BW, Mak CC, Ibanez M, Ghias A, Cahiwat J, Do L, Cho S, Nguyen J, Deshmukh V, Stewart J, Chen CW, Barroga C, Dellamary L, Kc SK, Phalen TJ, Hood J, Cha S, Yazici Y. The CLK inhibitor SM08502 induces anti-tumor activity and reduces Wnt pathway gene expression in gastrointestinal cancer models. Cancer Lett. 2020 Mar 31;473:186-197. doi: 10.1016/j.canlet.2019.09.009. Epub 2019 Sep 24. PMID 31560935